CLINICAL TRIAL: NCT06777966
Title: Effect of Preoperative Nebulized Versus Intravenous Tranexamic Acid on Surgical Field Quality in Patients Undergoing Endoscopic Sinus Surgeries: a Randomized Controlled Comparative Study
Brief Title: Nebulized Versus Intravenous Tranexamic Acid on Surgical Field Quality in Patients Undergoing Endoscopic Sinus Surgeries
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kareem Mohammed Assem Nawwar, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MD-206-2024
Record Dates: First submitted 2025-01-11; First posted 2025-01-16 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Nebulization; Intravenous; Surgical Field; Endoscopic Sinus Surgeries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebulized group (Active Comparator): patients will receive nebulized tranexamic acid
  Interventions: Drug: nebulized tranexamic acid
- Intravenous group (Active Comparator): patients will receive intravenous tranexamic acid
  Interventions: Drug: intravenous tranexamic acid

INTERVENTIONS:
Drug: nebulized tranexamic acid — patients will receive a preoperative nebulizer session of 500 mg of tranexamic acid. To ensure the blinding of the participating anesthetist and patient, patients in this group will receive an intravenous drip of 100 ml of 0.9% normal saline.
  Arms: Nebulized group
Drug: intravenous tranexamic acid — patients will receive a preoperative intravenous drip of TXA at a dose of 15 mg/kg in 100 ml of normal saline. To ensure blinding this group patients will receive 5 ml of 0.9% normal saline nebulizer session.
  Arms: Intravenous group

SUMMARY:
Intraoperative bleeding is one of the vital problems for anesthesiologists and surgeons, during endoscopic nasal surgery; where the surgical field is very limited and surrounded by vital structures. The tinniest amount of blood in such surgical field can obscure the anatomy and clog the tip of the endoscope, requiring repeated irrigations and suctioning; both of which have traumatic effects on the friable nasal mucosa. Anesthetic techniques to minimize bleeding during endoscopic nasal surgery are of primary importance for a safe and effective procedure, reducing operative time and shortening post-operative recovery.

Good surgical conditions could be achieved with systemic, topical, or regional anesthetic techniques. The use of topical and regional techniques has been gaining popularity in recent years as an alternative to the administration of heavy premedication, high narcotic doses, intravenous lignocaine, clonidine, calcium channel blockers, sodium nitroprusside, beta-adrenergic blockers, and magnesium sulfate, which may produce a lack of alertness, respiratory depression, hypoxia, nausea and vomiting, and delayed recovery.

Recent studies have shown that the use of tranexamic acid could be a safe and effective management option for hemostasis in a wide range of specialties. Tranexamic acid (TXA) is a synthetic lysine derivative that blocks the lysine binding site on plasminogen, thus inactivating its conversion to plasmin and hence attenuating its fibrinolysis effects. When given as a one-time operative systemic dose, it can reduce intraoperative surgical blood loss. More recently, it has been used in its nebulized or topical form to treat bleeding in anatomically sequestered areas. Its use has been described for epistaxis, cancer-related hemoptysis, and post-tonsillectomy bleeding. Though systemic doses of tranexamic acid have proven their efficiency in reducing intraoperative bleeding, other forms of administration have not been widely researched. The use of nebulized form is expected to provide a targeted route and localized effect with reduced systemic side effects. Adverse effects of systemic administration of tranexamic acid include seizures, nausea, vomiting, diarrhea, pulmonary embolism, deep vein thrombosis, anaphylaxis, and other visual disturbance.

The purpose of this study was to assess the effect of pre-emptive nebulized tranexamic acid versus intravenous tranexamic acid on endoscopic visualization and bleeding rate during endoscopic sinus surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years.
* American Society of Anesthesiologists (ASA) class I and II patients.
* Endoscopic sinus surgeries under general anesthesia.

Exclusion Criteria:

* Patient's refusal.
* American Society of Anesthesiologists (ASA) class III or IV patients.
* Underlying uncontrolled hypertension.
* Known history bleeding disorder.
* Patients on anticoagulant therapy.
* Allergy to any of the drugs utilized in this study.
* History of nonsteroidal anti-inflammatory drugs within 48 hours of scheduled surgery.
* Inadvertent intra-operative vascular injury.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-18 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The mean Wormald intraoperative surgical field grading | 5 hours
  The mean value of Wormald intraoperative surgical field grading throughout the intraoperative period, where 0 means no bleeding and 10 means severe bleeding with nasal cavity filling rapidly

SECONDARY OUTCOMES:
Total blood loss | 5 hours
  calculated by measuring the volume of the blood in the suction reservoir minus the normal saline used to wash the surgical field
Bleeding rate | 5 hours
  calculated as the total blood loss divided by the surgical time
Operation time | 5 hours
  Time starting from induction of anesthesia till completion of the surgical procedure
Postoperative complications | 24 hours
  nausea, vomiting, anaphylaxis, visual impairment, seizure, venous thromboembolism
postoperative nasal bleeding | 48 hours
  Incidence of postoperative nasal bleeding
postoperative intervention | 48 hours
  Incidence of the need for postoperative intervention to control nasal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Nevan M Abbas Elmekawy, M.D., Study Chair — Cairo University; Tamer M Khair, M.D., Study Director — Cairo University; Kareem MA Nawwar, M.D., Study Director — Cairo University; Nadia E M Gaballah, M.Sc., Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt